CLINICAL TRIAL: NCT00156234
Title: Training and Congestive Heart Failure
Brief Title: Skeletal Muscle Dysfunction in Heart Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ullevaal University Hospital (Other)
Collaborators: Norwegian Health Association (Other); Norwegian School of Sport Sciences (Other); The Research Council of Norway (Other); University of Oslo (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Educational/Counseling/Training
Other Study IDs: TRUST-001; Helse Øst; Helse og rehabilitering
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2005-09-12 (Estimated); Status verified 2005-09

CONDITIONS: Heart Failure, Congestive
MeSH Terms: conditions — Heart Failure

INTERVENTIONS:
Behavioral: One-knee extension ergometer

SUMMARY:
Patients suffering from congestive heart failure report reduced exercise capacity. This skeletal muscle dysfunction is also detectable when using small muscle groups which should not put any demand on the heart.

We hypothesize that congestive heart failure has systemic effects that causes the skeletal muscle dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Coronary Heart Failure
* Ejection fraction <35%
* NYHA 2-3
* Spirometry FEV1 > 80%

Exclusion Criteria:

* Cardiomyopathy
* Transplantation candidate
* Active malignancy
* Restraining skeletal-muscular disease
* Claudication in legs
* Hospitalized last 30 days due to acute ischemic episode
* Intravenous inotrope or vasodilatating drugs last 14 days prior to inclusion
* AMI last 8 weeks prior to inclusion
* Organized training last 4 months
* Smoking on daily basis last 4 months
* Creatinin < 150microliters/liter

Ages: 40 Years to 78 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45
Dates: Start 2005-03

CONTACTS AND LOCATIONS:
Overall Officials: Ole M Sejersted, Professor, Study Chair — Institute for Experimental Medical Research, Ullevaal University Hospital; Per Kristian B Lunde, Post Doc, Study Director — Institute for Experimental Medical Research, Ullevaal University Hospital; Ivar Sjaastad, Post Doc, Study Director — Institute for Experimental Medical Research, Ullevaal University Hospital; Jostein Hallen, Professor, Study Chair — Norwegian School of Sport Sciences; Morten Munkvik, Ph.D student, Principal Investigator — Institute for Experimental Medical Research, Ullevaal University Hospital; Tommy A Rehn, Vit.ass., Principal Investigator — Institute for Experimental Medical Research, Ullevaal University Hospital; Gunnar S Petersen, Ph.D student, Principal Investigator — Norwegian School of Sport Sciences
Locations (2):
- Norway (2):
  - Institute for Experimental Medical Research, Oslo, Oslo County
  - Norwegian School of Sport Sciences, Oslo, Oslo County

REFERENCES:
- [Derived] Munkvik M, Rehn TA, Slettalokken G, Hasic A, Hallen J, Sjaastad I, Sejersted OM, Lunde PK. Training effects on skeletal muscle calcium handling in human chronic heart failure. Med Sci Sports Exerc. 2010 May;42(5):847-55. doi: 10.1249/MSS.0b013e3181c29ec1. PMID 19996998